CLINICAL TRIAL: NCT05348148
Title: Camillian Saint Mary's Hospital Luodong
Brief Title: Comparison of the Effects for Lightening the Shiners Among Different Treatments for Rhinitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Camillians Saint Mary's Hospital Luodong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB109005
Record Dates: First submitted 2021-12-22; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Allergic Rhinitis; Vasomotor Rhinitis
Keywords: shiners; rhinitis
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Vasomotor; Rhinitis | interventions — levocetirizine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The independent researchers will carry out the digital image analyze.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral Levocetirizine (Active Comparator): Patients in Levocetirizine group will use oral antihistamine (Levocetirizine) only
  Interventions: Drug: Oral Levocetirizine
- Combined Intranasal Mometasone Furoate with oral Levocetirizine (Active Comparator): Patients in combined Intranasal Mometasone Furoate with oral Levocetirizineintranasal group will use combined intranasal corticosteroids (intranasal Mometasone Furoate) with oral antihistamine (Levocetirizine)
  Interventions: Drug: Combined Intranasal Mometasone Furoate with oral Levocetirizine
- Combined Intranasal Mometasone Furoate with oral Levocetirizine plus intranasal Oxymetazoline (Active Comparator): The other in combined Intranasal Mometasone Furoate with oral Levocetirizine plus intranasal Oxymetazoline group will use combined intranasal corticosteroids (intranasal Mometasone Furoate) with oral antihistamine (Levocetirizine) plus one-week intranasal decongestant (intranasal Oxymetazoline)
  Interventions: Drug: Combined Intranasal Mometasone Furoate with oral Levocetirizine plus intranasal Oxymetazoline

INTERVENTIONS:
Drug: Oral Levocetirizine — Patients will be randomly assigned into three groups. Patients in oral Levocetirizine group will use oral antihistamine only (Levocetirizine), another in combined Intranasal Mometasone Furoate with oral Levocetirizine group will use combined intranasal corticosteroids (intranasal Mometasone Furoate) with oral antihistamine (Levocetirizine), and the other in combined Intranasal Mometasone Furoate with oral Levocetirizine plus intranasal Oxymetazoline group will use combined intranasal corticosteroids (intranasal Mometasone Furoate) with oral antihistamine (Levocetirizine) plus one-week intranasal decongestant (intranasal Oxymetazoline).
  Digital images and the questionnaires, including PRQLQ, AdolRQLQ, and mini-RQLQ, of every participant will be taken at the beginning of the study. Further assessments will be taken at least 3 times, on the seventh day, fourteenth day, and twenty-eighth day after treatment.
  Arms: Oral Levocetirizine
Drug: Combined Intranasal Mometasone Furoate with oral Levocetirizine — Patients will be randomly assigned into three groups. Patients in oral Levocetirizine group will use oral antihistamine only (Levocetirizine), another in combined Intranasal Mometasone Furoate with oral Levocetirizine group will use combined intranasal corticosteroids (intranasal Mometasone Furoate) with oral antihistamine (Levocetirizine), and the other in combined Intranasal Mometasone Furoate with oral Levocetirizine plus intranasal Oxymetazoline group will use combined intranasal corticosteroids (intranasal Mometasone Furoate) with oral antihistamine (Levocetirizine) plus one-week intranasal decongestant (intranasal Oxymetazoline).
  Digital images and the questionnaires, including PRQLQ, AdolRQLQ, and mini-RQLQ, of every participant will be taken at the beginning of the study. Further assessments will be taken at least 3 times, on the seventh day, fourteenth day, and twenty-eighth day after treatment.
  Arms: Combined Intranasal Mometasone Furoate with oral Levocetirizine
Drug: Combined Intranasal Mometasone Furoate with oral Levocetirizine plus intranasal Oxymetazoline — Patients will be randomly assigned into three groups. Patients in oral Levocetirizine group will use oral antihistamine only (Levocetirizine), another in combined Intranasal Mometasone Furoate with oral Levocetirizine group will use combined intranasal corticosteroids (intranasal Mometasone Furoate) with oral antihistamine (Levocetirizine), and the other in combined Intranasal Mometasone Furoate with oral Levocetirizine plus intranasal Oxymetazoline group will use combined intranasal corticosteroids (intranasal Mometasone Furoate) with oral antihistamine (Levocetirizine) plus one-week intranasal decongestant (intranasal Oxymetazoline).
  Digital images and the questionnaires, including PRQLQ, AdolRQLQ, and mini-RQLQ, of every participant will be taken at the beginning of the study. Further assessments will be taken at least 3 times, on the seventh day, fourteenth day, and twenty-eighth day after treatment.
  Arms: Combined Intranasal Mometasone Furoate with oral Levocetirizine plus intranasal Oxymetazoline

SUMMARY:
Background: Shiners are caused when blood and other fluids accumulate in the infraorbital groove. It develops resulting from lots of problems. In patient with rhinitis, either allergic rhinitis or non-allergic rhinitis, shiners are believed to be caused by venous stasis resulting from nasal congestion. This study is aiming that comparison of the effectiveness of treatment of rhinitis (either allergic rhinitis or non-allergic rhinitis) to lighten not only the rhinitis but also the shiners. Randomized control studies.

Design: The investigators will recruit children (6-12 y/0), adolescent (13-18 y/o), or adults (19-65 y/o) with either allergic rhinitis or non-allergic rhinitis, and patients will be randomly assigned to groups (oral antihistamine, combined nasal corticosteroids with oral antihistamine, combined nasal corticosteroids with oral antihistamine plus nasal decongestant, combined nasal corticosteroids with oral antihistamine plus nasal irrigation, combined oral antihistamine with nasal irrigation, or nasal antihistamine only). Digital image will be recorded and analyzed to compare the change of shiners between before and after treatment for rhinitis. The clinical data were collected including patient's data, history, laboratory data, Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ), Adolescent Rhinoconjunctivitis Quality of Life Questionnaire (AdolRQLQ), or mini Rhinoconjunctivitis Quality of Life Questionnaire (mini-RQLQ), and medications. The primary outcome is to answer whether the levels of shiners can be alleviated by using therapies in patient with rhinitis. And the secondary outcome is to figure out which therapies work most effectively.

Keywords: allergic rhinitis, vasomotor rhinitis, shiners, nasal corticosteroids

DETAILED DESCRIPTION:
Background:

Shiners results from the accumulation of body fluid in the infraorbital groove. The physiology and pathology in children include nasal congestion, inﬂammation of nose and eyes, trauma to the nose or the forehead, facial surgery, or facial cancer. In patient with either allergic rhinitis or non-allergic rhinitis, nasal congestion arouses venous stasis, leading to the blue-gray to purple discoloration under the bilateral lower eyelids, called shiners. In patients with allergic rhinitis, allergic shiners, termed by Marks since 1954, have been regarded as a significant sign of allergic rhinitis generally.

In 2009, Chiang and members established a digital-analyzed tool to quantify allergic shiners, and the results demonstrated the darkness and the area values of allergic shiners correlate with the severity of allergic rhinitis.

A stepwise approach for the treatment of allergic rhinitis and non-allergic rhinitis is documented, including oral antihistamine, intranasal antihistamine, intranasal corticosteroids, intranasal decongestant, oral or intranasal leukotriene antagonist, as well as nasal irrigation, but the response of shiners after treatment, and the efficiency of the therapies to alleviate the shiners were unknown. In this study, the primary outcome is to answer whether the levels of shiners can be alleviated by using nasal therapies in patients with allergic rhinitis or non-allergic rhinitis. And the secondary outcome is to figure out which nasal therapies work most effectively.

Design:

The investigators will recruit children (6-12 years old), adolescent (13-18 years old), and adults (19-65 years old) with moderate to severe rhinitis, either allergic rhinitis or non-allergic rhinitis. Those with chronic rhinosinusitis, trauma to the forehead or nose, face surgery, malignancy, pregnancy, and respiratory tract infections or usage of medications for rhinitis within a week before beginning the study will be excluded. Study population will be classified into children, adolescent and adults according to the age.

This study will be divided into three stages. In the first stage, three kinds of therapies for rhinitis were compared. Patients will be randomly assigned into three groups. Patients in group 1 will use oral antihistamine only, another in group 2 will use combined intranasal corticosteroids with oral antihistamine, and the other in group 3 will use combined intranasal corticosteroids with oral antihistamine plus one-week intranasal decongestant. In the second stage, three kinds of therapies will be compared, including combined intranasal corticosteroids and oral antihistamine, combined intranasal corticosteroids and oral antihistamine plus nasal irrigation, and oral antihistamine plus nasal irrigation. The third stage will compare oral antihistamine only, combined intranasal corticosteroids with oral antihistamine, and intranasal antihistamine. The estimated sample size was 50 cases in each groups, and total 150 cases in each population and total 450 cases in each stage. Patients will be randomized by a randomization table. Minimization will be performed when over 100 cases in each population and in each stage.

A standardized digital photograph of every participant will be recorded and further analyzed to compare the change of shiners between before and after treatment for rhinitis. The clinical data will be collected including patient's data, history, laboratory data, Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) of every children, Adolescent Rhinoconjunctivitis Quality of Life Questionnaire (AdolRQLQ) of every adolescent, or mini Rhinoconjunctivitis Quality of Life Questionnaire (mini-RQLQ) of every adult, and medications.

Digital images and the questionnaires, including PRQLQ, AdolRQLQ, and mini-RQLQ, of every participant will be taken at the beginning of the study. Further assessments will be taken at least 3 times, on the seventh day, fourteenth day, and twenty-eighth day after treatment.

The detail method to take a standardized digital photography, and analyze digital image were described in the previous study. Briefly, in order to standardize both the size and color of the photographs, a color checker used as a reference was set in front of the every participant's chin. Pixel, the elemental unit of digital image, was calculated in each photographs. After completing preprocess in every digital sample, the investigators converted the intensity value of each pixel into the gray level, then measured the gray-level mean values in the infraorbital groove (Sm) and cheek (Cm), respectively. Darkness (D) was equal to Cm-Sm. The blacker a shiner appeared, the bigger the darkness value was. Shiner's area value was figured out by sampling the curve of each lower eyes. The investigators translated the value from pixels to square centimeters, and finally normalized by body surface area to gain the parameter A (in square centimeters per square meter) represented as the area value of shiner.

The independent researchers will carry out the digital image analyze.

The primary outcome is to answer whether the levels of shiners can be alleviated by using therapies in patient with rhinitis. And the secondary outcome is to figure out which therapies work most effectively.

Statistical analysis The investigators compared the categorical variables between the two groups using the Pearson's Chi square test. The investigators compared the continuous variables between the two groups using Mann-Whitney U test. The correlation between two parameters was analyzed by Pearson correlation test. The investigators used paired samples t-test and/or multiple regression analysis to what kind of treatment was more effective to alleviate the shiners with/without improvement of rhinitis. To account for correlation among repeated measures from the same patient, the study was analyzed with the usage of linear generalized estimating equations. A p value < 0.05 was considered statistically significant. All statistical analyses were performed with International Business Machines Corporation Statistical Product and Service Solutions statistical software (version 20.0.0, IBM Corp., Armonk, NY).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderate to severe rhinitis, either allergic rhinitis or non-allergic rhinitis.

Exclusion Criteria:

* Chronic rhinosinusitis
* Trauma to the forehead or nose
* Face surgery
* Malignancy
* Pregnancy
* Respiratory tract infections within a week before beginning the study
* Usage of medications for rhinitis within a week before beginning the study

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2032-03-31 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
alleviating darkness of shiners | Change from baseline darkness of shiners at 1 week after treatment.
  Change from baseline of the darkness of shiners at 1 week after treatment.
alleviating darkness of shiners | Change from baseline darkness of shiners at 2 weeks after treatment.
  Change from baseline of the darkness of shiners at 2 week after treatment.
alleviating darkness of shiners | Change from baseline darkness of shiners at 4 weeks after treatment.
  Change from baseline of the darkness of shiners at 4 week after treatment.
alleviating area value of shiners | Change from baseline area value of shiners at 1 week after treatment.
  Change from baseline of the area value of shiners at 1 week after treatment.
alleviating area value of shiners | Change from baseline area value of shiners at 2 week after treatment.
  Change from baseline of the area value of shiners at 2 week after treatment.
alleviating area value of shiners | Change from baseline area value of shiners at 4 week after treatment.
  Change from baseline of the area value of shiners at 4 week after treatment.

SECONDARY OUTCOMES:
alleviating darkness of shiners among groups | Change from baseline darkness of shiners at 1 week after treatment.
  Change from baseline of the darkness of shiners at 1 week after treatment among groups (including oral Levocetirizine group, combined Intranasal Mometasone Furoate with oral Levocetirizine group, and combined Intranasal Mometasone Furoate with oral Levocetirizine plus intranasal Oxymetazoline group).
alleviating darkness of shiners among groups | Change from baseline darkness of shiners at 2 week after treatment.
  Change from baseline of the darkness of shiners at 2 week after treatment among groups (including oral Levocetirizine group, combined Intranasal Mometasone Furoate with oral Levocetirizine group, and combined Intranasal Mometasone Furoate with oral Levocetirizine plus intranasal Oxymetazoline group).
alleviating darkness of shiners among groups | Change from baseline darkness of shiners at 4 week after treatment.
  Change from baseline of the darkness of shiners at 4 week after treatment among groups (including oral Levocetirizine group, combined Intranasal Mometasone Furoate with oral Levocetirizine group, and combined Intranasal Mometasone Furoate with oral Levocetirizine plus intranasal Oxymetazoline group).
alleviating area value of shiners among groups | Change from baseline area value of shiners at 1 week after treatment.
  Change from baseline of the area value of shiners at 1 week after treatment among groups (including oral Levocetirizine group, combined Intranasal Mometasone Furoate with oral Levocetirizine group, and combined Intranasal Mometasone Furoate with oral Levocetirizine plus intranasal Oxymetazoline group).
alleviating area value of shiners among groups | Change from baseline area value of shiners at 2 week after treatment.
  Change from baseline of the area value of shiners at 2 week after treatment among groups (including oral Levocetirizine group, combined Intranasal Mometasone Furoate with oral Levocetirizine group, and combined Intranasal Mometasone Furoate with oral Levocetirizine plus intranasal Oxymetazoline group).
alleviating area value of shiners among groups | Change from baseline area value of shiners at 4 week after treatment.
  Change from baseline of the area value of shiners at 4 week after treatment among groups (including oral Levocetirizine group, combined Intranasal Mometasone Furoate with oral Levocetirizine group, and combined Intranasal Mometasone Furoate with oral Levocetirizine plus intranasal Oxymetazoline group).

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Tsung Yang, Principal Investigator — Camillian Saint Mary's Hospital Luodong
Locations (1):
- Camillian Saint Mary's Hospital Luodong, Luodong, Yilan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marks MB. Allergic shiners. Dark circles under the eyes in children. Clin Pediatr (Phila). 1966 Nov;5(11):655-8. doi: 10.1177/000992286600501106. No abstract available. PMID 5926923
- [Result] Goren SB. Eye disorders: common ocular injuries: assessing the severity. Postgrad Med. 1975 Dec;58(7):99-102. doi: 10.1080/00325481.1975.11714225. PMID 1197147
- [Result] Chuan MT, Tsai TF, Wu MC, Wong TH. Atrophic pigmented dermatofibrosarcoma presenting as infraorbital hyperpigmentation. Dermatology. 1997;194(1):65-7. doi: 10.1159/000246061. PMID 9031796
- [Result] Lai L, Casale TB, Stokes J. Pediatric allergic rhinitis: treatment. Immunol Allergy Clin North Am. 2005 May;25(2):283-99, vi. doi: 10.1016/j.iac.2005.02.003. PMID 15878456
- [Result] Marks MB. Photo of eye depression. In: Vaughan WT, Black JR, editors. Practice of allergy. Philadelphia: C.V. Mosby Co; 1954. p. 1023
- [Result] MARKS MB. Nasal allergy in childhood. Observations in the South Florida area. Ann Allergy. 1960 Oct;18:1110-6. No abstract available. PMID 13766957
- [Result] Marks MB. Significance of discoloration in the lower orbitopalpebral grooves in allergic children (allergic shiners). Ann Allergy 1963;21:26-32.
- [Result] Berger WE. Allergic rhinitis in children : diagnosis and management strategies. Paediatr Drugs. 2004;6(4):233-50. doi: 10.2165/00148581-200406040-00003. PMID 15339201
- [Result] Quillen DM, Feller DB. Diagnosing rhinitis: allergic vs. nonallergic. Am Fam Physician. 2006 May 1;73(9):1583-90. PMID 16719251
- [Result] Prenner BM, Schenkel E. Allergic rhinitis: treatment based on patient profiles. Am J Med. 2006 Mar;119(3):230-7. doi: 10.1016/j.amjmed.2005.06.015. PMID 16490466
- [Result] Chen CH, Lin YT, Wen CY, Wang LC, Lin KH, Chiu SH, Yang YH, Lee JH, Chiang BL. Quantitative assessment of allergic shiners in children with allergic rhinitis. J Allergy Clin Immunol. 2009 Mar;123(3):665-71, 671.e1-6. doi: 10.1016/j.jaci.2008.12.1108. PMID 19281911
- [Result] Bousquet J, Van Cauwenberge P, Khaltaev N; Aria Workshop Group; World Health Organization. Allergic rhinitis and its impact on asthma. J Allergy Clin Immunol. 2001 Nov;108(5 Suppl):S147-334. doi: 10.1067/mai.2001.118891. No abstract available. PMID 11707753
- [Result] Sur DKC, Plesa ML. Chronic Nonallergic Rhinitis. Am Fam Physician. 2018 Aug 1;98(3):171-176. PMID 30215894
- [Result] Scadding GK, Kariyawasam HH, Scadding G, Mirakian R, Buckley RJ, Dixon T, Durham SR, Farooque S, Jones N, Leech S, Nasser SM, Powell R, Roberts G, Rotiroti G, Simpson A, Smith H, Clark AT. BSACI guideline for the diagnosis and management of allergic and non-allergic rhinitis (Revised Edition 2017; First edition 2007). Clin Exp Allergy. 2017 Jul;47(7):856-889. doi: 10.1111/cea.12953. PMID 30239057
- [Result] Agnihotri NT, McGrath KG. Allergic and nonallergic rhinitis. Allergy Asthma Proc. 2019 Nov 1;40(6):376-379. doi: 10.2500/aap.2019.40.4251. PMID 31690374
- [Result] Wise SK, Lin SY, Toskala E, Orlandi RR, Akdis CA, Alt JA, Azar A, Baroody FM, Bachert C, Canonica GW, Chacko T, Cingi C, Ciprandi G, Corey J, Cox LS, Creticos PS, Custovic A, Damask C, DeConde A, DelGaudio JM, Ebert CS, Eloy JA, Flanagan CE, Fokkens WJ, Franzese C, Gosepath J, Halderman A, Hamilton RG, Hoffman HJ, Hohlfeld JM, Houser SM, Hwang PH, Incorvaia C, Jarvis D, Khalid AN, Kilpelainen M, Kingdom TT, Krouse H, Larenas-Linnemann D, Laury AM, Lee SE, Levy JM, Luong AU, Marple BF, McCoul ED, McMains KC, Melen E, Mims JW, Moscato G, Mullol J, Nelson HS, Patadia M, Pawankar R, Pfaar O, Platt MP, Reisacher W, Rondon C, Rudmik L, Ryan M, Sastre J, Schlosser RJ, Settipane RA, Sharma HP, Sheikh A, Smith TL, Tantilipikorn P, Tversky JR, Veling MC, Wang Y, Westman M, Wickman M, Zacharek M. International Consensus Statement on Allergy and Rhinology: Allergic Rhinitis. Int Forum Allergy Rhinol. 2018 Feb;8(2):108-352. doi: 10.1002/alr.22073. PMID 29438602
- [Result] Brozek JL, Bousquet J, Agache I, Agarwal A, Bachert C, Bosnic-Anticevich S, Brignardello-Petersen R, Canonica GW, Casale T, Chavannes NH, Correia de Sousa J, Cruz AA, Cuello-Garcia CA, Demoly P, Dykewicz M, Etxeandia-Ikobaltzeta I, Florez ID, Fokkens W, Fonseca J, Hellings PW, Klimek L, Kowalski S, Kuna P, Laisaar KT, Larenas-Linnemann DE, Lodrup Carlsen KC, Manning PJ, Meltzer E, Mullol J, Muraro A, O'Hehir R, Ohta K, Panzner P, Papadopoulos N, Park HS, Passalacqua G, Pawankar R, Price D, Riva JJ, Roldan Y, Ryan D, Sadeghirad B, Samolinski B, Schmid-Grendelmeier P, Sheikh A, Togias A, Valero A, Valiulis A, Valovirta E, Ventresca M, Wallace D, Waserman S, Wickman M, Wiercioch W, Yepes-Nunez JJ, Zhang L, Zhang Y, Zidarn M, Zuberbier T, Schunemann HJ. Allergic Rhinitis and its Impact on Asthma (ARIA) guidelines-2016 revision. J Allergy Clin Immunol. 2017 Oct;140(4):950-958. doi: 10.1016/j.jaci.2017.03.050. Epub 2017 Jun 8. PMID 28602936
- [Result] Wheatley LM, Togias A. Clinical practice. Allergic rhinitis. N Engl J Med. 2015 Jan 29;372(5):456-63. doi: 10.1056/NEJMcp1412282. PMID 25629743
- [Result] Seidman MD, Gurgel RK, Lin SY, Schwartz SR, Baroody FM, Bonner JR, Dawson DE, Dykewicz MS, Hackell JM, Han JK, Ishman SL, Krouse HJ, Malekzadeh S, Mims JW, Omole FS, Reddy WD, Wallace DV, Walsh SA, Warren BE, Wilson MN, Nnacheta LC; Guideline Otolaryngology Development Group. AAO-HNSF. Clinical practice guideline: Allergic rhinitis. Otolaryngol Head Neck Surg. 2015 Feb;152(1 Suppl):S1-43. doi: 10.1177/0194599814561600. PMID 25644617
- [Result] Sur DK, Plesa ML. Treatment of Allergic Rhinitis. Am Fam Physician. 2015 Dec 1;92(11):985-92. PMID 26760413
- [Result] Piromchai P, Puvatanond C, Kirtsreesakul V, Chaiyasate S, Thanaviratananich S. Effectiveness of nasal irrigation devices: a Thai multicentre survey. PeerJ. 2019 May 27;7:e7000. doi: 10.7717/peerj.7000. eCollection 2019. PMID 31179187
- [Result] Chong LY, Head K, Hopkins C, Philpott C, Glew S, Scadding G, Burton MJ, Schilder AG. Saline irrigation for chronic rhinosinusitis. Cochrane Database Syst Rev. 2016 Apr 26;4(4):CD011995. doi: 10.1002/14651858.CD011995.pub2. PMID 27115216
- [Result] Juniper EF, Howland WC, Roberts NB, Thompson AK, King DR. Measuring quality of life in children with rhinoconjunctivitis. J Allergy Clin Immunol. 1998 Feb;101(2 Pt 1):163-70. doi: 10.1016/s0091-6749(98)70380-x. PMID 9500748
- [Result] Juniper EF, Guyatt GH, Dolovich J. Assessment of quality of life in adolescents with allergic rhinoconjunctivitis: development and testing of a questionnaire for clinical trials. J Allergy Clin Immunol. 1994 Feb;93(2):413-23. doi: 10.1016/0091-6749(94)90349-2. PMID 8120268
- [Result] Juniper EF, Thompson AK, Ferrie PJ, Roberts JN. Development and validation of the mini Rhinoconjunctivitis Quality of Life Questionnaire. Clin Exp Allergy. 2000 Jan;30(1):132-40. doi: 10.1046/j.1365-2222.2000.00668.x. PMID 10606940